CLINICAL TRIAL: NCT02496546
Title: An Explorative Trial Evaluating the Effect of LEO 32731 Cream 20 mg/g in Adults With Mild to Moderate Atopic Dermatitis (AD)
Brief Title: An Explorative Trial Evaluating the Effect of LEO 32731 Cream in Adults With Mild to Moderate Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0108-1082; 2014-000519-15 (EudraCT Number)
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 32731 cream (Experimental): Topical application
  Interventions: Drug: LEO 32731 cream
- LEO 32731 cream vehicle (Placebo Comparator): Topical application
  Interventions: Drug: LEO 32731 cream vehicle

INTERVENTIONS:
Drug: LEO 32731 cream — Applied for 3 weeks
  Arms: LEO 32731 cream
Drug: LEO 32731 cream vehicle — Applied for 3 weeks
  Arms: LEO 32731 cream vehicle

SUMMARY:
The aim of this trial is to assess the efficacy of LEO 32731 cream 20 mg/g compared with LEO 32731 cream vehicle in adults with mild to moderate AD after 3 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Following verbal and written information about the trial, subjects must provide informed consent documented by signing the Informed Consent Form (ICF) prior to any trial related procedures being carried out
* Subject with Atopic Dermatitis (AD) as defined by Hanifin and Rajka criteria and with mild to moderate disease severity (IGA 2 or 3) as assessed by a dermatologically trained investigator (and confirmed by a board certified dermatologist before or at visit 1)
* Two symmetrically located and comparable Entire Treatment Areas (ETAs) of 20 - 50 cm2 each, i.e. on the same body region (left and right part) and of the same size (complete AD lesion or part of an AD lesion); Total Sign Score (TSS) of at least 5 on both ETAs; difference in TSS not greater than 2 between the two ETAs; sign score for erythema ≥ 2 on both ETAs; difference in Investigator´s Treatment Area assessment of disease severity not greater than 1 between the 2 ETAs

Exclusion Criteria:

* Any condition in the treatment areas that in the opinion of the investigator could interfere with clinical assessments, e.g. acne, infection, rash (other than Atopic Dermatitis), sunburn, hyper- or hypopigmentation, scars

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Total sign score at end of treatment on entire treatment area | 3 weeks
  Total sign score is defined as the sum of severity scores (4-point scale) of the Individual Sign Scores (erythema, edema/papulation, oozing/crusting, excoriations, lichenification and dryness) for each area

SECONDARY OUTCOMES:
Total sign score on limited treatment area on entire treatment area during trial | 3 week
Investigator's treatment area assessment of disease severity on entire treatment area during trial | 3 weeks
Subject's treatment area assessment of disease severity on entire treatment area during trial | 3 weeks
Subject's assessment of itching on entire treatment area during trial | 3 weeks
Transepidermal water loss during trial | 3 weeks
Individual signs score on entire treatment during trial | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Proinnovera GmbH, Center of Dermatology Excellence, Münster, Germany